CLINICAL TRIAL: NCT02469454
Title: Effect of the Immediately Postpartum Insertion of the Etonogestrel Releasing Implant on Infant Growth and Development
Brief Title: Effect of t of the Etonogestrel Releasing Implant on Infant Growth and Development
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Carolina Sales Vieira, MD, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: ENG-implant-02
Record Dates: First submitted 2015-06-09; First posted 2015-06-11 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Contraception; Newborn; Child Development; Growth
Keywords: etonogestrel-implant; newborn; growth; Child Development

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- early insertion (Experimental): Postpartum women into whom the etonogestrel-releasing contraceptive implant (Implanon®, N.V. Organon, Oss, Netherlands) will be inserted in the first 48 h postpartum. The ENG implant will be inserted subdermally in the non-dominant arm of volunteers upon local anesthesia with 2% lidocaine with vasoconstrictor, according to the manufacturer's instructions.
  Interventions: Drug: early insertion
- conventional insertion (Active Comparator): Postpartum women into whom the etonogestrel-releasing contraceptive implant (Implanon®, N.V. Organon, Oss, Netherlands) will be inserted after 6 week of the delivery. The ENG implant will be inserted subdermally in the non-dominant arm of volunteers upon local anesthesia with 2% lidocaine with vasoconstrictor, according to the manufacturer's instructions.
  Interventions: Drug: conventional insertion

INTERVENTIONS:
Drug: early insertion — Postpartum women into whom the etonogestrel-releasing contraceptive implant (Implanon®, N.V. Organon, Oss, Netherlands) will be inserted in the first 48 h postpartum.
  Arms: early insertion
Drug: conventional insertion — Postpartum women into whom the etonogestrel-releasing contraceptive implant (Implanon®, N.V. Organon, Oss, Netherlands) will be inserted in the first 6 week of delivery.
  Arms: conventional insertion

SUMMARY:
This study aims to assess whether there is change in the growth and development of newborns whose mothers will have a etonogestrel (ENG) releasing implant inserted in the first 24 to 48 hours of delivery compared with those with standard implant insertion (6 week postpartum).

ELIGIBILITY:
Inclusion Criteria:

* Women who desire to use the ENG implant as a contraceptive method and desire to breastfeed her newborn for ate least 3 months;
* With no contraindication to breastfeeding, whose newborn is healthy, without malformations, born at term (gestational age ≥ 37 weeks), with appropriate weight for gestational age and with normal sucking ability

Exclusion Criteria:

* Tobacco smokers, drug addicts or alcoholics;
* Women with educational levels lower than 5 years;
* Women with clinical conditions considered category 3 and 4 for implant use by the WHO;
* Women with histories of psychiatric illness;
* Women using medications that could alter the concentration of ENG,
* Women with known allergies to the local anesthetic lidocaine (used to place the implant);
* Women who wanted to keep their cyclic menstrual bleeding

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2015-06; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
neonatal growth | 12 months

SECONDARY OUTCOMES:
child development | 12 months
  Child development will be evaluated by Bayley III Scale

CONTACTS AND LOCATIONS:
Overall Officials: Carolina S Vieira, MD, PhD, Principal Investigator — Sao Paulo University
Locations (1):
- Clinical Hospital of Sao Paulo University, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Nadai MN, Martins Linhares MB, de Lima Rodrigues Sisdeli JC, de Melo Pereira do Carmo LS, Braga GC, Ferreira LS, Quintana SM, Vieira CS. Effects of the immediate postpartum insertion of the etonogestrel implant on the development of breastfed infants: Results from a randomized controlled trial. Int J Gynaecol Obstet. 2025 Dec;171(3):1223-1230. doi: 10.1002/ijgo.70291. Epub 2025 Jun 9. PMID 40488538
- [Derived] Vieira CS, de Nadai MN, de Melo Pereira do Carmo LS, Braga GC, Infante BF, Stifani BM, Ferriani RA, Quintana SM. Timing of postpartum etonogestrel-releasing implant insertion and bleeding patterns, weight change, 12-month continuation and satisfaction rates: a randomized controlled trial. Contraception. 2019 Oct;100(4):258-263. doi: 10.1016/j.contraception.2019.05.007. Epub 2019 May 27. PMID 31145885
- [Derived] Carmo LSMP, Braga GC, Ferriani RA, Quintana SM, Vieira CS. Timing of Etonogestrel-Releasing Implants and Growth of Breastfed Infants: A Randomized Controlled Trial. Obstet Gynecol. 2017 Jul;130(1):100-107. doi: 10.1097/AOG.0000000000002092. PMID 28594758